CLINICAL TRIAL: NCT04410952
Title: Bleeding Control in Type-C Pelvic Ring Fractures Using the Pelvic C-clamp vs. the Pelvic Binder for Emergency Stabilization - a Matched Pair Analysis From the German Pelvic Registry
Brief Title: Pelvic Binder vs. Pelvic C-clamp for Bleeding Control
Status: Completed | Type: Observational
Sponsor: BG Trauma Center Tuebingen (Other)
Responsible Party: Principal Investigator, Markus Küper, PD Dr. med., BG Trauma Center Tuebingen
Other Study IDs: 002
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Pelvic Ring Fracture; Pelvic Bleeding; Polytrauma
Keywords: Pelvic binder; Pelvic C-clamp; Pelvic ring fracture; Fatal pelvic bleeging; Emergency stabilization
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- no EES: Patients with a Type-C pelvic ring fracture who underwent no external emergency stabilization (EES) for the posterior pelvic ring
- Pelvic binder: Patients with a Type-C pelvic ring fracture who received a pelvic binder for emergency stabilization of the posterior pelvic ring
- Pelvic C-clamp: Patients with a Type-C pelvic ring fracture who received a pelvic C-clamp for emergency stabilization of the posterior pelvic ring

SUMMARY:
Pelvic ring fractures carry a high risk for severe bleeding. Expecially bleeding from the posterior ring might result in a fatal course. Different types of external emergency stabilization (EES) are available for the posterior pelvic ring, namely the non-invasive pelvic binder or the invasive pelvic c-clamp. Which stabilization technique is superior, has not been investigated yet.

DETAILED DESCRIPTION:
Severe bleeding is the major cause of death in unstable pelvic ring fractures. Therefore, a quick and efficient emergency stabilization and bleeding control is inevitable. The pelvic C-clamp and the pelvic binder are efficient tools for temporary bleeding control, especially for the posterior pelvic ring. However, whether these disadvantages make up for a more efficient bleeding control, still needs to be discussed in the guidelines of the emergency management of pelvic ring fractures.

Patients with a type-C pelvic ring fracture were identified from the German Pelvic Registry (GPR). The patients were divided into three groups of 40 patients: 1. group without emergency stabilization, 2. group treated with pelvic binder and 3. group treated with pelvic C-clamp. The patients were matched according to the following parameters: age, gender, initial RR and HB level. The complication rates and mortality rates were compared between the groups, especially regarding bleeding control, as measured by the amount of transfused blood products. Furthermore, the subjective efficacy of the treatment was assessed. Finally, the time until established bleeding control was compared.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for data acquisition in the German Pelvic Registry
* Pelvic ring fracture Type C (AO/OTA)
* ISS (Abdomen) >8

Exclusion Criteria:

* Acetabular fracture
* Pelvic ring fracture Type A/B (AO/OTA)
* ISS (Abdomen) <9

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a Type-C pelvic ring fracture and an abdominal ISS >8 are identified from the German Pelvic Registry.
  Cases in which the external emergency stabilization was not specified were left included. The remaining cases were divided into the different treatment groups:
  1. Patients who received no external emergency stabilization.
  2. Patients who were treated with a pelvic binder.
  3. Patients who were treated with a C-clamp.
  Age, gender, the initial HB level and the initial blood pressure were used to match the cases of the three groups.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Need for transfusion | 24 hours
  Number of transfused units of packed red blood cells
Time until emergency stabilization | 6 hours
  The time until emergency stabilization device is placed in minutes

SECONDARY OUTCOMES:
Mortality rate | 6 months
  The rate of deaths due to fatal bleeding
Length of hospital stay | 6 months
  Duration of the inpatient treatment in days
Complication rate | 6 months
  The rate of overall complications

CONTACTS AND LOCATIONS:
Overall Officials: Markus A. Küper, MD, Principal Investigator — BG Trauma Center Tübingen
Locations (1):
- BG Trauma Center, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF